CLINICAL TRIAL: NCT02695823
Title: Incidence of Intracranial Hypertension During Liver Transplantation Estimated by Non-invasive Ultrasound Methods.
Acronym: TOH-HTIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL15_0483
Record Dates: First submitted 2016-02-11; First posted 2016-03-01 (Estimated); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Liver Transplantation
Keywords: intracranial hypertension; liver transplantation; transcranial Doppler; optic nerve sheath diameter
MeSH Terms: conditions — Intracranial Hypertension | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients undergoing liver transplantation (Experimental)
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — Ultrasound measurements of the optic nerve sheath diameter and intracranial Doppler, at 4 time points during surgery (incision, anhepatic phase + 30 min, declamping + 5 min, declamping + 30 min), and at day 1 and day 5 after surgery, to detect presence of intracranial hypertension.
  Search of any neurological complication during the 5 postoperative days.

SUMMARY:
Acute or chronic liver failure (fulminant hepatitis or advanced cirrhosis) disrupts brain physiology. Beyond classical hepatic encephalopathy, intracranial hypertension may occur.During liver transplantation (LT) surgery, many factors can lead to cerebral assault. In addition, intracranial hypertension measured with invasive methods has been described in certain phases of LT, especially at the time of reperfusion.

The invasive monitoring of the intracranial pressure is not used in these patients, due to a high risk of infection and bleeding. The non-invasive monitoring of intracranial pressure has been widely developed in recent years : transcranial doppler and recently ultrasound of the optic nerve sheath (ONSD) allow an effective detection of intracranial hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years
* Patients who underwent orthotopic liver transplantation
* Patients who have received clear information and not opposed to participate in the study
* Patients affiliated to a social security scheme or similar
* Patients not undergoing a measure of legal protection

Exclusion Criteria:

* Opposition to participation in the study
* Patients < 18 years
* Pregnant women or breastfeeding
* Deprived of individual liberty
* Non-affiliated to a social security scheme
* Known ophthalmic pathology: untreated cataracts, glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2015-12-09 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Measure of the optic nerve sheath diameter during surgery. | at incision
  A value of the optic nerve sheath diameter (averaged over 2 measures) greater than 5.7 mm will be considered pathological, indicating the strong likelihood of intracranial hypertension (PPV near 100% for an intracranial pressure > 25 cmh2o in the literature) The optic nerve sheath diameter will be measured by ultrasonography, in accordance with existing protocols: Use probe 7.5 Mhz in 2D mode, patient supine dorsi, implementation of ultrasound gel on the closed eyelid, search for the optimal window 3mm, optic nerve sheath diameter measurement behind the retina using an electronic cursor along an axis perpendicular to the optic nerve. 2 measurements per side (sagittal and transverse plane) averaged. Values> 5.7mm are deemed pathological.
Measure of the optic nerve sheath diameter during surgery. | at anhepatic phase + 30 min
  A value of the optic nerve sheath diameter (averaged over 2 measures) greater than 5.7 mm will be considered pathological, indicating the strong likelihood of intracranial hypertension (PPV near 100% for an intracranial pressure > 25 cmh2o in the literature) The optic nerve sheath diameter will be measured by ultrasonography, in accordance with existing protocols: Use probe 7.5 Mhz in 2D mode, patient supine dorsi, implementation of ultrasound gel on the closed eyelid, search for the optimal window 3mm, optic nerve sheath diameter measurement behind the retina using an electronic cursor along an axis perpendicular to the optic nerve. 2 measurements per side (sagittal and transverse plane) averaged. Values> 5.7mm are deemed pathological.
Measure of the optic nerve sheath diameter during surgery. | at declamping + 5 min
  A value of the optic nerve sheath diameter (averaged over 2 measures) greater than 5.7 mm will be considered pathological, indicating the strong likelihood of intracranial hypertension (PPV near 100% for an intracranial pressure > 25 cmh2o in the literature) The optic nerve sheath diameter will be measured by ultrasonography, in accordance with existing protocols: Use probe 7.5 Mhz in 2D mode, patient supine dorsi, implementation of ultrasound gel on the closed eyelid, search for the optimal window 3mm, optic nerve sheath diameter measurement behind the retina using an electronic cursor along an axis perpendicular to the optic nerve. 2 measurements per side (sagittal and transverse plane) averaged. Values> 5.7mm are deemed pathological.
Measure of the optic nerve sheath diameter during surgery. | at declamping + 30 min
  A value of the optic nerve sheath diameter (averaged over 2 measures) greater than 5.7 mm will be considered pathological, indicating the strong likelihood of intracranial hypertension (PPV near 100% for an intracranial pressure > 25 cmh2o in the literature) The optic nerve sheath diameter will be measured by ultrasonography, in accordance with existing protocols: Use probe 7.5 Mhz in 2D mode, patient supine dorsi, implementation of ultrasound gel on the closed eyelid, search for the optimal window 3mm, optic nerve sheath diameter measurement behind the retina using an electronic cursor along an axis perpendicular to the optic nerve. 2 measurements per side (sagittal and transverse plane) averaged. Values> 5.7mm are deemed pathological.

SECONDARY OUTCOMES:
Measurement of intracranial hypertension with transcranial Doppler during surgery. | at incision
  Diastolic velocity value of less than 20 cm s-1 and a pulsatility index greater than 1.4 will be considered pathological, indicating a high probability of intracranial hypertension.
  The transcranial Doppler measurements are performed according to the existing protocols: use of a cardiac probe 2 Mhz, positioned temporal window, the circle of Willis color Doppler tracking then collecting the Doppler signal of the middle cerebral artery in Doppler pulsed with the insonation angle as small as possible to a depth between 40 and 60 mm. Measuring systolic, diastolic and mean velocity )Vs, Vd, Vm) and calculating the pulsatility Index (PI) bilaterally. PI values of> 1.4 and Vd <20 cm s-1 will be considered pathological.
Measurement of intracranial hypertension with transcranial Doppler during surgery. | at anhepatic phase + 30 min
  Diastolic velocity value of less than 20 cm s-1 and a pulsatility index greater than 1.4 will be considered pathological, indicating a high probability of intracranial hypertension.
  The transcranial Doppler measurements are performed according to the existing protocols: use of a cardiac probe 2 Mhz, positioned temporal window, the circle of Willis color Doppler tracking then collecting the Doppler signal of the middle cerebral artery in Doppler pulsed with the insonation angle as small as possible to a depth between 40 and 60 mm. Measuring systolic, diastolic and mean velocity )Vs, Vd, Vm) and calculating the pulsatility Index (PI) bilaterally. PI values of> 1.4 and Vd <20 cm s-1 will be considered pathological.
Measurement of intracranial hypertension with transcranial Doppler during surgery. | at declamping + 5 min
  Diastolic velocity value of less than 20 cm s-1 and a pulsatility index greater than 1.4 will be considered pathological, indicating a high probability of intracranial hypertension.
  The transcranial Doppler measurements are performed according to the existing protocols: use of a cardiac probe 2 Mhz, positioned temporal window, the circle of Willis color Doppler tracking then collecting the Doppler signal of the middle cerebral artery in Doppler pulsed with the insonation angle as small as possible to a depth between 40 and 60 mm. Measuring systolic, diastolic and mean velocity )Vs, Vd, Vm) and calculating the pulsatility Index (PI) bilaterally. PI values of> 1.4 and Vd <20 cm s-1 will be considered pathological.
Measurement of intracranial hypertension with transcranial Doppler during surgery. | at declamping + 30 min
  Diastolic velocity value of less than 20 cm s-1 and a pulsatility index greater than 1.4 will be considered pathological, indicating a high probability of intracranial hypertension.
  The transcranial Doppler measurements are performed according to the existing protocols: use of a cardiac probe 2 Mhz, positioned temporal window, the circle of Willis color Doppler tracking then collecting the Doppler signal of the middle cerebral artery in Doppler pulsed with the insonation angle as small as possible to a depth between 40 and 60 mm. Measuring systolic, diastolic and mean velocity )Vs, Vd, Vm) and calculating the pulsatility Index (PI) bilaterally. PI values of> 1.4 and Vd <20 cm s-1 will be considered pathological.
Measurement of intracranial hypertension with transcranial Doppler | at 1 day after surgery.
  we use the same methods and the same thresholds as those used during surgery (primary outcome measure, and measure1 of secondary outcome measure)
Measure of the optic nerve sheath diameter after surgery. | at 1 day after surgery.
  we use the same methods and the same thresholds as those used during surgery (primary outcome measure, and measure1 of secondary outcome measure)
Measurement of intracranial hypertension with transcranial Doppler | at 5 days after surgery.
  we use the same methods and the same thresholds as those used during surgery (primary outcome measure, and measure1 of secondary outcome measure)
Measure of the optic nerve sheath diameter after surgery. | at 5 days after surgery.
  we use the same methods and the same thresholds as those used during surgery (primary outcome measure, and measure1 of secondary outcome measure)
The early appearance of neurological complications after surgery. | During the 5 days following surgery
  A monitoring with simultaneous collection of clinical, biological and ultrasound parameters, will be done. Neurological complications after surgery will be defined by the presence of at least one of the following criteria: Glasgow score < 14 in a non-sedated patient, behavioral disorders, agitation (evaluation according to the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) score), epilepsy, imaging or MRI scan. Pathological evolved compared to the preoperative including hemorrhagic or thrombotic cardiovascular event. Various confounding factors will be considered (serum sodium, serum tacrolimus, serum magnesium, ammonia, sedatives).

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu GAZON, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Département d'anesthésie réanimation, Lyon, France